CLINICAL TRIAL: NCT00744705
Title: Normative Database of the Retinal Nerve Fiber Layer Thickness Measured by the Cirrus HD OCT in Asians
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Gong Je Seong, Yonsei University College of Medicine
Other Study IDs: 3-2008-0076-3
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2008-09-01 (Estimated); Status verified 2008-08

CONDITIONS: Glaucoma
Keywords: Retinal nerve fiber layer; Glaucoma; Myopia
MeSH Terms: conditions — Glaucoma; Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Normal subjects who received routine health check-up in a comprehensive medical testing center

SUMMARY:
The normal range of retinal nerve fiber layer thickness might be different between Asians and Caucasians. However, the recently developed imaging device such as the Cirrus HD OCT includes only the Caucasian data. So, the investigators want to find its normal range of in Asians.

DETAILED DESCRIPTION:
Characteristics of various ocular parameters are influenced by race. Because the retinal nerve fiber layer (RNFL) thickness is crucial in detecting early glaucomatous changes, its normal range is also important. Even though the normal range of RNFL thickness might be different according to race, the recently developed imaging device such as the Cirrus HD OCT includes only the Caucasian data. In the present study, we want to measure the RNFL thickness using the Cirrus HD OCT in normal Asian eyes and to determine its normal range in Asians.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects
* Good quality of the OCT images (signal intensity > 8)

Exclusion Criteria:

* Any ocular history
* DM

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal subjects who recieved a regular medical check-up in a comprehensive medical testing center of our institute
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-11 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Retinal nerve fiber layer thickness | when the OCT images are taking

SECONDARY OUTCOMES:
Refractive errors | when the OCT images are taking
Intraocular pressure | when the OCT images are taking

CONTACTS AND LOCATIONS:
Overall Officials: Gong Je Seong, MD, PhD, Study Chair — Yonsei University
Locations (1):
- Yongdong Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea